CLINICAL TRIAL: NCT05081895
Title: Ventilation and Perfusion in the Respiratory System
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Alex Pearce, Principal Investigator, University of California, San Diego
Other Study IDs: 210285
Record Dates: First submitted 2021-09-09; First posted 2021-10-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Failure; Respiratory Distress Syndrome, Adult; Critical Illness; Pulmonary Disease; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Critical Illness; Lung Diseases; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Respiratory failure
  Interventions: Device: Electrical Impedance tomography; Other: Lung mechanics and gas exchange

INTERVENTIONS:
Device: Electrical Impedance tomography — Patients will be monitored with electrical impedance tomography during routine care with special attention to effects of neuromuscular blockade and postural changes.
Other: Lung mechanics and gas exchange — Patient lung mechanics and gas exchange will be monitored during routine clinical care, with specific attention to postural changes and use of neuromuscular blockade.

SUMMARY:
Respiratory failure occurs when the lung fails to perform one or both of its roles in gas exchange; oxygenation and/or ventilation. Presentations of respiratory failure can be mild requiring supplemental oxygen via nasal cannula to more severe requiring invasive mechanical ventilation as see in acute respiratory distress syndrome (ARDS).It is important to provide supportive care through noninvasive respiratory support devices but also to minimize risk associated with those supportive devices such as ventilator induced lung injury (VILI) and/or patient self-inflicted lung injury (P-SILI). Central to risk minimization is decreasing mechanical stress and strain and optimizing transpulmonary pressure or the distending pressure across the lung, minimizing overdistention and collapse. Patient positioning impacts ventilation/perfusion and transpulmonary pressure. Electrical impedance tomography (EIT) is an emerging technology that offers a noninvasive, real-time, radiation free method to assess distribution of ventilation at the bedside. The investigators plan to obtain observational data regarding distribution of ventilation during routine standard of care in the ICU, with special emphasis on postural changes and effects of neuromuscular blockade, to provide insight into ventilation/perfusion matching, lung mechanics in respiratory failure, other pulmonary pathological processes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* admitted to UC San Diego La Jolla or Hillcrest Campus Intensive Care Units
* Patient requiring supplemental oxygen (including but no limited to nasal cannula, high flow devices, noninvasive positive pressure ventilation or mechanical ventilation

Exclusion Criteria:

* <18 years
* Chest wall, anatomical, physical abnormalities, skin integrity issues precluding placement of electrode belt in direct contact with skin
* Patient is too unstable to position the belt/electrodes or tolerate head of bed changes
* Confirmed or suspected intracranial bleed, stroke, edema
* Active implants (i.e. implantable electronic devices such as pacemakers, cardioverter defibrillators, neurostimulators) or if device compatibility is in doubt
* Pregnant or lactating patients as safety and efficacy for use of EIT in such cases has not been verified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human subjects admitted to the UC San Diego La Jolla Campus and Hillcrest Campus Intensive Care Units who are admitted with a pathologic condition requiring supplemental oxygen (including but not limited to nasal cannula, high flow devices), noninvasive positive pressure ventilation, mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Distribution of ventilation | change from baseline at 15 minutes and 1 hour
  Regional ventilation distribution differences measured through electrical impedance tomography (EIT)

SECONDARY OUTCOMES:
Lung mechanics | Baseline, then at 15 minutes and 1 hour
  Lung compliance
Oxygenation | Up to 48 hours
  Oxygen saturation measured by pulse oximetry (SpO2) and fraction of inspired oxygen (FiO2) as well as arterial blood gas partial pressure of oxygen (PaO2). Results will be reported as either PaO2/FiO2 ratio or SpO2/FiO2 ratio (depending on availability of arterial blood gas measurements)
Blood Gas Partial Pressure of Carbon Dioxide (PaCO2) (mmHg) | Up to 48 hours
  Partial pressure of carbon dioxide (PaCO2) (mmHg)
Blood Gas pH | Up to 48 hours
  Blood Gas pH

OTHER OUTCOMES:
In-hospital Mortality | Up to 28 days
  Mortality at 28 days after study enrollment
ICU Mortality | Up to 28 days
  ICU Mortality
Ventilator-free days | Up to 28 days
  Ventilator-free days
Ventilator associated pneumonia | Up to 28 days
  Incidence of ventilator associated pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Alex Pearce, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests for IPD will be considered by the investigators